CLINICAL TRIAL: NCT04359953
Title: Efficacy of Hydroxychloroquine, Telmisartan and Azithromycin on the Survival of Hospitalized Elderly Patients With COVID-19: a Randomized, Multicenter, Adaptative Study
Brief Title: Efficacy of Hydroxychloroquine, Telmisartan and Azithromycin on the Survival of Hospitalized Elderly Patients With COVID-19
Acronym: COVID-Aging
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: difficulty in recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7747
Record Dates: First submitted 2020-04-17; First posted 2020-04-24 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: COVID-19 Infection
Keywords: COVID-19; Elderly; Therapeutic study
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; Azithromycin; Telmisartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hydroxychloroquine (Experimental): Patient will take 200mg of Hydroxychloroquine twice a day during 14 days
  Interventions: Drug: Hydroxychloroquine
- Azithromycin (Experimental): Patient will take 250mg of Azithromycin twice a day during 14 days
  Interventions: Drug: Azithromycin
- Telmisartan (Experimental): Patient will take 40mg of Telmisartan twice a day during 14 days
  Interventions: Drug: Telmisartan
- Usual Care (No Intervention): No intervention

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine 2 x per day during 14 days
  Arms: Hydroxychloroquine
Drug: Azithromycin — Azithromycin 2 x per day during 14 days
  Arms: Azithromycin
Drug: Telmisartan — Telmisartan 2 x per day during 14 days
  Arms: Telmisartan

SUMMARY:
In November 2019, Wuhan city in China, became the center of an outbreak of pneumonia due to a novel coronavirus SARS-CoV-2, which disease was named coronavirus disease 2019 (COVID19) in February, 2020. The COVID19 is much more dangerous for people over 60 with a death rate of 3.6% after 60, 8.0% after 70 and 14.8% after 80 -and according to our Italian colleagues over 20% after 90- against 2.3% in the general population. The elderly patients who died most often had multiple comorbidities and in particular: cardiovascular disease (10.5% mortality), diabetes (7.3%), chronic respiratory disease (6.3%) and hypertension (6%). These elderly patients with COVID19 are therefore very fragile and require treatment that fights the virus but is also adapted to their state of health and age. Most of current therapeutic trials worldwide exclude people aged over 75 years, which is precisely the age group affected by COVID19. We therefore propose to carry out a therapeutic trial specific to the elderly with drugs at doses that are bearable for these patients. Using the WHO, clinicaltrial, pubmed and the Chinese CCDC/CHCTR websites to find the better drugs adapted to elderly people, we decided after concertation between infectiologists and geriatricians to do a four arms clinical trial during two weeks twice a day: Hydroxychloroquine 200mg, Telmisartan 40mg, Azithromycin 250mg and standard care. We therefore hypothesize that one or more of these treatments may have a beneficial effect in controlling COVID19, without major and repeated side effects in elderly patients.

DETAILED DESCRIPTION:
In the absence of a validated treatment, any patient over 75 years -or demented above 60- of age arriving in one of our hospital centres with a COVID19 infection objectified by RT-PCR will be offered this therapeutic trial. Patients will be randomized. During their hospitalization, they will be closely monitored clinically. It means daily evaluation of temperature, pulse, respiratory rate, blood pressure, need for oxygen therapy and general clinical examination. The lung severity scale and WHO scale will be done daily. Any side effects of any kind, in particular serious side effects will be reported within 24 hours on the electronic CRF. RT-PCR with search for SARS-Cov-2 will be evaluated at D0, D7 and D14. A blood sample will be taken at D0, D7 and D14 with blood count, CRP and biobanking. Functional scales (ADL, confusion scale, walking) will be evaluated every 3 days. If death occurs, the precise circumstances and time of death will be transmitted, as well as the precise origin of death: only COVID19 or other associated disease (bacterial infection, heart failure, kidney failure, etc...).

Symptomatic treatment will be at the discretion of the clinician, but will be recorded in the eCRF, particularly in relation to the use of corticosteroids or other immunomodulators.

The study will consist of 1600 patients over 75 years of age (or above 60 demented) with COVID19 requiring hospitalization, equally divided into four groups with the following treatment during two weeks for each arm:

* Hydroxychloroquine 200mg twice a day
* Azithromycin 250 mg twice a day
* Telmisartan 40mg twice a day
* Standard care

The choice of these three drugs was done considering the benefit-risk balance, i.e. by choosing drugs with few side effects but high potential for elderly people (including severe renal insufficiency). Hydroxychloroquine was chosen because 1. This drug was demonstrated to be potent and more potent than Chloroquine at inhibiting SARS-CoV-2 in vitro. An unpublished clinical trial with 100 patients showing superiority of chloroquine compared to placebo with improvement of lung image findings, promotion a virus-negative conversion and shortening the disease course . An open-label non randomized clinical trial with 42 patients showing a faster reduction of the virus in the Hydroxychloroquine treated group. Azithromycin was associated in the previous trial with Hydroxychloroquine with positive results on RT-PCR. Recently bioinformatic analysis conclude to SARS-CoV-2 protease inhibition with Macrolides. Moreover macrolides are known to have immunomodulatory effects, which could be of interest in the context of hyperinflammation. Telmisartan is an angiotensin 2 AT1 receptor antagonist. COVID19 use ACE2 as a receptor, a modulator of the activity of different angiotensin. The COVID19-ACE2 interaction increases the activity of angiotensin and thus increases the activity of the AT1 receptor, that results in increased pulmonary vascular permeability and therefore contributes to lung injury. Thus Telmisartan could be a protector against lung injury due to Sars-Cov-2, inhibiting AT1 receptor.

The expected benefits are multiple thanks to this original project:

* 1. There is a research emergency. No drug has been shown to be really effective against COVID19 and even less in the elderly, so therapeutic trials are needed.
* 2. If one of these 3 drugs turns out to be positive, it could even be taken at a very early stage, for example as a result of a recent contagion, in elderly population at high risk of death.
* 3. If one of the three treatments was positive, the cost-effectiveness would be very favorable compared to other treatments currently being tested. This could benefit a larger population, particularly in developing countries where COVID19 is arriving.
* 4. This trial will be evolutionary, i.e. we will be able to add a treatment arm if a new molecule that is potentially effective in the elderly appears.

ELIGIBILITY:
Inclusion Criteria:

* Subject Male or female age ≥ 75, or ≥ 60 if dementia
* Subject infected with COVID 19 (confirmed by RT-PCR SARS-CoV-2 detectable less than 5 days old and clinical picture)
* Clinical manifestation of COVID 19 requiring hospitalization:

pneumopathy and/or upper airway infection and/or respiratory distress, confusion and/or encephalopathy and/or signs of encephalitis, walking disorders with ataxia and/or falls, digestive problem (diarrhea and/or vomiting)

* Subject affiliated to a social health insurance scheme
* Subject capable of understanding the objectives and risks of the research and of giving dated and signed informed consent, or agreement given by a trusted person, guardian or trustee.
* Subject who has been informed of the results of the prior medical examination

Exclusion Criteria:

* Patients with a negative RT-PCR SARS-CoV-2 result
* Patients with COVID19 pneumopathy requiring resuscitative breathing support
* Porphyria
* Kaliemia 3.5 mmol/l and 5.5 mmol/l
* Any reason why patient follow-up would be impossible during the study period
* Patient on Sartan (Telmisartan, Candesartan, Valsartan, etc...), another antihypertensive, Hydroxychloroquine or Chloroquine, or macrolides (Azithromycin, Clarythromycyin...) within the last 24 hours.
* Patient with a contraindication to one of the treatments proposed in the study
* Contraindication Hydroxychloroquine: citalopram, escitalopram, hydroxyzine, domperidone, piperaquine, QT prolongation (>470ms for men and >480 ms for women), retinopathy, hypersensitivity to the active substances or to one of the excipients, known deficit in G6PD
* Contraindication Azithromycin: combination with ergot derivatives, combination with colchicine, patients at risk of developing cardiac arrhythmia (diagnosis of QTc interval prolongation (>470ms for men and >480 ms for women), severe hepatic impairment,severe cholestase, history of allergy to macrolides or any of the excipients used in this study, end-stage renal failure with a glomerular filtration rate (DFG) - 15 ml/min, patients with malignant hemopathies who have undergone an allograft of hematopoietic stem cells
* Contraindication Telmisartan: Combination with drugs containing aliskiren, severe hepatic impairment, biliary obstruction, hypersensitivity to the active substance or to any of the excipients used in this study.
* Subject under safeguard of justice

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-04-25 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Two-weeks survival rate | Day 14

SECONDARY OUTCOMES:
Rate of undetectable RT-PCR of SARS-CoV-2 | Day 7
Rate of undetectable RT-PCR of SARS-CoV-2 | Day 14
Rate of death | Day 28
Hypotension | Day 7
Hypotension | Day 14
Hypothermia and hyperthermia | Day 7
Hypothermia and hyperthermia | Day 14
Pneumonia severity according to WHO | Day 7
Pneumonia severity according to PSI (Hung et al 2017) | Day 7
Pneumonia severity according to WHO | Day 14
Pneumonia severity according to PSI (Hung et al 2017) | Day 14
Rate of no cough | Day 7
Rate of no cough | Day 14
Rate of no dyspnea | Day 7
Rate of no dyspnea | Day 14
Rate of no fever | Day 7
Rate of no fever | Day 14
Rate of no requiring supplemental oxygen | Day 7
Rate of no requiring supplemental oxygen | Day 14
Rate of SARS-Cov-2 undetectable | Day 7
Rate of SARS-Cov-2 undetectable | Day 14
Recovery time | Day 28
Critical admission rate | Day 28
Mechanical ventilation rate | Day 28
Changes in Activity of Daily Living (ADL) Activity of Daily Living) | Day 13
Changes in Activity of Daily Living IADL (Instrumental Activity of Daily Living) | Day 13
The number and dose of added corticosteroids, immonumodulators or immunosuppressants | Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric BLANC, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- CHU de Strasbourg, Strasbourg, France